CLINICAL TRIAL: NCT02130635
Title: A Double-Blind (Sponsor Unblind), Placebo Controlled, Randomised, Parallel Group Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Doses of GSK2269557 Administered as a Dry Powder to COPD Patients and Assessment of Dose Response Using Sputum Biomarkers
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Dose-Response Relationship of Multiple Doses of GSK2269557 Administered as a Dry Powder to Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115119
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: PI3Kd; Pharmacodynamics; dry powder inhaler; GSK2269557; safety; COPD subjects
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nemiralisib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Part A: GSK2269557 1000 MCG (Experimental): Subjects will receive 2 inhalations (2 x GSK2269557 500 mcg = total dose of 1000 mcg GSK2269557) 30 seconds apart, once daily for 14 consecutive days
  Interventions: Drug: GSK2269557 500 MCG
- Part A: PLACEBO (Placebo Comparator): Subjects will receive 2 inhalations of placebo once daily for 14 consecutive days
  Interventions: Drug: PLACEBO
- Part B: GSK2269557 100 MCG (Experimental): Subjects will receive 4 inhalations (1 x GSK2269557 100 mcg and 3 x Placebo = total dose of 100 mcg GSK2269557) 30 seconds apart, once daily for 14 consecutive days
  Interventions: Drug: GSK2269557 100 MCG; Drug: PLACEBO
- Part B: GSK2269557 200 MCG (Experimental): Subjects will receive 4 inhalations (2 x GSK2269557 100 mcg and 2 x Placebo = total dose of 200 mcg GSK2269557) 30 seconds apart, once daily for 14 consecutive days
  Interventions: Drug: GSK2269557 100 MCG; Drug: PLACEBO
- Part B: GSK2269557 500 MCG (Experimental): Subjects will receive 4 inhalations (1 x GSK2269557 500 mcg and 3 x Placebo = total dose of 500 mcg GSK2269557) 30 seconds apart, once daily for 14 consecutive days, once daily for 14 consecutive days
  Interventions: Drug: GSK2269557 500 MCG; Drug: PLACEBO
- Part B: GSK2269557 700 MCG (Experimental): Subjects will receive 4 inhalations (1 x GSK2269557 500 mcg, 2 x GSK2269557 100 mcg and 1 x Placebo = total dose of 700 mcg GSK2269557) 30 seconds apart, once daily for 14 consecutive days
  Interventions: Drug: GSK2269557 100 MCG; Drug: GSK2269557 500 MCG; Drug: PLACEBO
- Part B: GSK2269557 1000 MCG (Experimental): Subjects will receive 4 inhalations (2 x GSK2269557 100 mcg and 2 x Placebo = total dose of 1000 mcg GSK2269557) 30 seconds apart, once daily for 14 consecutive days
  Interventions: Drug: GSK2269557 500 MCG; Drug: PLACEBO
- Part B: GSK2269557 2000 MCG (Experimental): Subjects will receive 4 inhalations (2 x GSK2269557 100 mcg and 2 x Placebo = total dose of 2000 mcg GSK2269557) 30 seconds apart, once daily for 14 consecutive days
  Interventions: Drug: GSK2269557 500 MCG
- Part B: PLACEBO (Placebo Comparator): Subjects will receive 4 inhalations of placebo once daily for 14 consecutive days
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: GSK2269557 100 MCG — 100 mcg of GSK2269557 blended with lactose per blister administered using a dry powder inhaler device
  Arms: Part B: GSK2269557 100 MCG; Part B: GSK2269557 200 MCG; Part B: GSK2269557 700 MCG
Drug: GSK2269557 500 MCG — 500 mcg of GSK2269557 blended with lactose per blister administered using a dry powder inhaler device
  Arms: Part A: GSK2269557 1000 MCG; Part B: GSK2269557 1000 MCG; Part B: GSK2269557 2000 MCG; Part B: GSK2269557 500 MCG; Part B: GSK2269557 700 MCG
Drug: PLACEBO — Lactose administered using a matching dry powder inhaler device
  Arms: Part A: PLACEBO; Part B: GSK2269557 100 MCG; Part B: GSK2269557 1000 MCG; Part B: GSK2269557 200 MCG; Part B: GSK2269557 500 MCG; Part B: GSK2269557 700 MCG; Part B: PLACEBO

SUMMARY:
This is a randomised, double-blind, placebo controlled, parallel group study to evaluate the safety, tolerability, pharmacokinetics and dose response of multiple doses of GSK2269557 administered as a dry powder in COPD subjects. Pharmacodynamic effects on biomarkers will also be assessed. This study will have two parts. In Part A, subjects will be randomized to active or placebo treatment in a 3:1 ratio and in Part B, to placebo or one of the six doses of active treatment in an equal ratio. A sufficient number of COPD subjects (male and female of non-child bearing potential) will be screened to ensure that approximately 30 subjects are enrolled and at least 20 evaluable subjects are obtained for Part A and approximately 35 subjects will be enrolled for Part B. In both the parts, subjects will receive study treatment once daily for 14 consecutive days. Placebo control will be included for a valid evaluation of adverse events attributable to treatment versus those independent of treatment.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a confirmed and established diagnosis of COPD, as defined by the Global Initiative for Chronic Obstructive lung Disease (GOLD) guidelines.
* Male or female of non-child bearing potential between 40 and 75 years of age inclusive, at the time of signing the informed consent.
* The subject has a post-bronchodilator [400 microgram (mcg) salbutamol] Maximal amount of air FEV1/FVC <0.7 and FEV1 >=40% to <=80% of predicted (Predictions should be according to the European Community of Coal and Steel (ECCS) equations).
* Subject is a smoker or an ex-smoker with a smoking history of at least 10 pack years (pack years = (cigarettes per day smoked/20) x number of years smoked)).
* The subject is able to produce >100 milligram (mg) of sputum at screening.
* Body weight >=45 kilogram (kg) and body mass index (BMI) within the range 17 - 32 kg/square meter (m^2) (inclusive).
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, hysterectomy, salpingo-oophrectomy or oophrectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-International units (MIU)/millilitre (mL) and estradiol < 40 picogram (pg)/mL (<147 picomole(pmol)/Liter [L]) is confirmatory]. [Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.]; or has only same-sex partners, when this is her preferred and usual lifestyle.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until the follow-up visit.
* Based on averaged QTcF values of triplicate ECGs obtained over a brief recording period (e.g. 5 minutes): QTcF <450 millisecond (msec); or QTcF<480 msec in subjects with right bundle branch block.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included if the investigator [in consultation with the Glaxosmithkline (GSK) medical monitor if required] documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome, asymptomatic gallstones and cholecystectomy).
* Subjects who have a past or current medical condition or diseases that are not well controlled and, which as judged by the Investigator, may affect subject safety or influence the outcome of the study. (Note: Patients with adequately treated and well controlled concurrent medical conditions (e.g. hypertension) are permitted to be entered into the study).
* Subject has a diagnosis of active tuberculosis, lung cancer, clinically overt bronchiectasis, pulmonary fibrosis, asthma or any other respiratory condition that might, in the opinion of the Investigator, compromise the safety of the subject or affect the interpretation of the results.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >28 units for males or >21 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components (such as lactose) thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* A positive test for Human immunodeficiency virus (HIV) antibody - tested according to local policies.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include cannabinoids, amphetamines, barbiturates, cocaine and opiates. The detection of drugs (e.g. benzodiazepines, opiates) taken for a legitimate medical purpose would not necessarily be an exclusion to study participation. The detection of alcohol would not be an exclusion at screening but would need to be negative pre-dose and during the study.
* A positive pre-study Hepatitis B surface antigen (HBs-Ag) or positive total hepatitis B core antibody (anti-HBc IgM) or positive Hepatitis C antibody result within 3 months of screening.
* Pregnant females as determined by positive urine human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Subject has poorly controlled or unstable COPD, defined as the occurrence of any of the following: Either: acute worsening of COPD (an exacerbation) that is managed by the subject at home requiring treatment with corticosteroids and/or antibiotics in the 4 weeks prior to the screening visit; or more than two exacerbations in the previous 2 months prior to the screening visit that required a course of oral corticosteroids and/or antibiotics, or for which the subject was hospitalised.
* Subject has had a respiratory tract infection treated with antibiotics in the 4 weeks prior to first dose.
* Subject requires regular treatment with oral corticosteroids or has received oral or parenteral corticosteroids within 4 weeks of screening.
* Vulnerable subject (e.g., person kept in detention).
* The subject is not able to understand and communicate in German or native language.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2015-08-18 (Actual); Study Completion 2015-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Germany (2):
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was comprised of two parts. In Part A, participants were randomized to active or placebo treatment in a 3:1 ratio and in Part B, to placebo or one of the six doses of active treatment in an equal ratio. Each part comprised a separate sample of participants.
Groups:
- Part A: Placebo: Participants received 2 inhalations of matching placebo once daily for 14 consecutive days.
- Part A: GSK2269577 1000 µg: Participants received repeat doses of GSK2269557 1000 micrograms (µg) (2 inhalations of 500 µg each from a single device) administered as a dry powder inhalation, once daily for 14 consecutive days.
- Part B: Placebo: Participants received four inhalations of matching placebo (from four inhalation devices) once daily for 14 consecutive days.
- Part B: GSK2269577 100 µg: Participants received repeat doses of GSK2269557 100 µg administered as a dry powder inhalation, once daily for 14 consecutive days. To maintain blinding, the total dose was delivered through four inhalation devices, each device containing either GSK2269557 100 µg or placebo.
- Part B: GSK2269577 200 µg: Participants received repeat doses of GSK2269557 200 µg administered as a dry powder inhalation, once daily for 14 consecutive days. To maintain blinding, the total dose was delivered through four inhalation devices, each device containing either GSK2269557 100 µg or placebo.
- Part B: GSK2269577 500 µg: Participants received repeat doses of GSK2269557 500 µg administered as a dry powder inhalation, once daily for 14 consecutive days. To maintain blinding, the total dose was delivered through four inhalation devices, each device containing either GSK2269557 500 µg or placebo.
- Part B: GSK2269577 700 µg: Participants received repeat doses of GSK2269557 700 µg administered as a dry powder inhalation, once daily for 14 consecutive days. To maintain blinding, the total dose was delivered through four inhalation devices, each device containing GSK2269557 100 µg, 500 µg, or placebo.
- Part B: GSK2269577 1000 µg: Participants received repeat doses of GSK2269557 1000 µg administered as a dry powder inhalation, once daily for 14 consecutive days. To maintain blinding, the total dose was delivered through four inhalation devices, each device containing either GSK2269557 500 µg or placebo.
- Part B: GSK2269577 2000 µg: Participants received repeat doses of GSK2269557 2000 µg administered as a dry powder inhalation, once daily for 14 consecutive days. To maintain blinding, the total dose was delivered through four inhalation devices, each device containing GSK2269557 500 µg.
Period: Part A-Safety and Tolerability
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Started | 7 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B-Dose-Response Relationship
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Started | 0 | 0 | 5 | 5 | 5 | 5 | 6 | 5 | 5
Completed | 0 | 0 | 5 | 5 | 5 | 5 | 6 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg | Total
Number analyzed (Participants) | 7 | 21 | 5 | 5 | 5 | 5 | 6 | 5 | 5 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] — Data provided for Part A Population: N=28
  Years
    number analyzed (Participants) | 7 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28
    (all) | 65.1 (5.81) | 60.5 (6.68) |  |  |  |  |  |  |  | 61.7 (6.68)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Data for Part B is presented. Population: N=36
  Years
    number analyzed (Participants) | 0 | 0 | 5 | 5 | 5 | 5 | 6 | 5 | 5 | 36
    (all) |  |  | 64.4 (4.45) | 61.6 (4.56) | 62.2 (8.23) | 65.4 (5.81) | 64.7 (7.26) | 62.4 (9.24) | 62.4 (6.43) | 63.3 (6.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 2 | 4 | 1 | 0 | 3 | 3 | 3 | 24
  Male | 6 | 14 | 3 | 1 | 4 | 5 | 3 | 2 | 2 | 40
Race/Ethnicity, Customized [Number; unit: Participants]
  White-White/Caucasian/European Heritage | 7 | 21 | 5 | 5 | 5 | 5 | 6 | 5 | 5 | 64

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With at Least One Non-serious Adverse Event (AE), Serious Adverse Event (SAE), or Drug-related Adverse Event
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, associated with liver injury and impaired liver function defined as alanine aminotransferase >=3 x upper limit of normal (ULN), and total bilirubin >=2 x ULN or international normalized ratio >1.5. AEs were classified as potentially drug-related, based on the investigator's judgment. Refer to the general AE/SAE module for a list of AEs and SAEs.
Time Frame: From the start of study treatment until follow-up (assessed for approximately 19 days)
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
Participants
  At least one AE | 2 | 9
  At least one SAE | 0 | 1
  At least one drug-related AE | 2 | 6

2. Primary Outcome: Part A: Change From Baseline in Counts of White Blood Cells (WBC), Total Neutrophils (Total Absolute Neutrophil Count [ANC]), Lymphocytes, Monocytes, Eosinophils, Basophils, and Platelets at the Indicated Time Points
Description: Blood samples were collected for measurement for the indicated tests. Baseline is Day 1 pre-dose. Change from Baseline at any post-dose visit was calculated as the post-dose visit value minus the Baseline value. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
10^9 cells per liter (GI/L)
  WBC; Day 7/Day 8, pre-dose | -0.736 (0.937) | -0.080 (1.387)
  WBC; Day 14, 24 h post dose | -0.140 (1.220) | -0.510 (0.947)
  Total ANC; Day 7/Day 8, pre-dose | -0.664 (0.624) | -0.363 (1.342)
  Total ANC; Day 14, 24 h post dose | -0.153 (0.887) | -0.547 (0.977)
  Lymphocytes; Day 7/Day 8, pre-dose | -0.033 (0.321) | 0.172 (0.597)
  Lymphocytes; Day 14, 24 h post dose | -0.049 (0.197) | 0.030 (0.245)
  Monocytes; Day 7/Day 8, pre-dose | -0.036 (0.074) | 0.046 (0.149)
  Monocytes; Day 14, 24 h post dose | 0.039 (0.178) | -0.022 (0.116)
  Eosinophils; Day 7/Day 8, pre-dose | -0.006 (0.051) | 0.032 (0.074)
  Eosinophils; Day 14, 24 h post dose | 0.001 (0.085) | 0.010 (0.075)
  Basophils; Day 7/Day 8, pre-dose | -0.001 (0.006) | 0.006 (0.015)
  Basophils; Day 14, 24 h post dose | -0.003 (0.013) | 0.002 (0.018)
  Platelets; Day 7/Day 8, pre-dose | 1.6 (20.58) | 17.9 (36.44)
  Platelets; Day 14, 24 h post dose | 14.7 (21.80) | 23.5 (37.43)

3. Primary Outcome: Part A: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) at the Indicated Time Points
Description: Blood samples were collected for measurement for the indicated tests. Baseline is Day 1 pre-dose. MCHC is one of the red blood cell (RBC) indices. Change from Baseline at any post-dose visit was calculated as the post-dose visit value minus the Baseline value. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 h post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams/Liter (g/L)
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
Grams/Liter (g/L)
  Hemoglobin; Day 7/Day 8, pre-dose | -1.3 (6.63) | 1.6 (4.17)
  Hemoglobin; Day 14, 24 h post dose | 0.3 (6.97) | 1.0 (4.12)
  MCHC; Day 7/Day 8, pre-dose | -5.3 (7.32) | -2.2 (4.54)
  MCHC; Day 14, 24 h post dose | -8.4 (4.39) | -2.4 (6.45)

4. Primary Outcome: Part A: Change From Baseline in Hematocrit at the Indicated Time Points
Description: as for outcome 2
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
Ratio
  Hematocrit; Day 7/Day 8, pre-dose | 0.003 (0.023) | 0.007 (0.013)
  Hematocrit; Day 14, 24 h post dose | 0.011 (0.019) | 0.006 (0.016)

5. Primary Outcome: Part A: Change From Baseline in Counts of RBCs and Reticulocytes at the Indicated Time Points
Description: as for outcome 2
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/Liter (TI/L)
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
10^12 cells/Liter (TI/L)
  RBCs; Day 7/Day 8, pre-dose | 0.023 (0.230) | 0.060 (0.141)
  RBCs; Day 14, 24 h post dose | 0.119 (0.201) | 0.063 (0.160)
  Reticulocytes; Day 7/Day 8, pre-dose | 0.005 (0.014) | 0.003 (0.009)
  Reticulocytes; Day 14, 24 h post dose | 0.009 (0.014) | 0.003 (0.010)

6. Primary Outcome: Part A: Change From Baseline in Mean Corpuscle Hemoglobin (MCH) at the Indicated Time Points
Description: Blood samples were collected for measurement for the indicated tests. Baseline is Day 1 pre-dose. MCH is one of the red blood cell indices. Change from Baseline at any post-dose visit was calculated as the post-dose visit value minus the Baseline value. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms (pg)
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
Picograms (pg)
  MCH; Day 7/Day 8, pre-dose | -0.46 (0.602) | -0.06 (0.440)
  MCH; Day 14, 24 h post dose | -0.76 (0.586) | -0.23 (0.593)

7. Primary Outcome: Part A: Change From Baseline in Mean Corpuscle Volume (MCV) at the Indicated Time Points
Description: Blood samples were collected for measurement for the indicated tests. Baseline is Day 1 pre-dose. MCV is one of the RBC indices. Change from Baseline at any post-dose visit was calculated as the post-dose visit value minus the Baseline value. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliters (fL)
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
Femtoliters (fL)
  MCV; Day 7/Day 8, pre-dose | 0.11 (0.687) | 0.43 (0.697)
  MCV; Day 14, 24 h post dose | 0.07 (0.848) | -0.03 (1.193)

8. Primary Outcome: Part A: Change From Baseline in Albumin and Total Protein at the Indicated Time Points
Description: as for outcome 2
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
g/L
  Albumin; Day 7/Day 8, pre-dose | 0.56 (2.230) | 0.80 (1.576)
  Albumin; Day 14, 24 h post doseTotal protein; Day | 0.53 (2.379) | 0.52 (2.004)
  Total protein; Day 7/Day 8, pre-dose | 0.56 (3.619) | 1.28 (2.599)
  Total protein; Day 14, 24 h post dose | 0.84 (3.887) | 1.15 (2.606)

9. Primary Outcome: Part A: Change From Baseline in Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), and Gamma Glutamyl Transferase (GGT) at the Indicated Time Points
Description: as for outcome 2
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
International Units per Liter (IU/L)
  ALT; Day 7/Day 8, pre-dose | 2.46 (2.585) | -0.61 (2.208)
  ALT; Day 14, 24 h post dose | 1.51 (2.667) | -0.40 (4.117)
  ALP; Day 7/Day 8, pre-dose | -0.64 (6.937) | 1.14 (8.586)
  ALP; Day 14, 24 h post dose | -2.23 (6.522) | -0.21 (9.785)
  AST; Day 7/Day 8, pre-dose | 3.14 (7.674) | -1.03 (3.081)
  AST; Day 14, 24 h post dose | 1.83 (4.750) | -0.71 (2.592)
  GGT; Day 7/Day 8, pre-dose | -0.91 (2.203) | 0.11 (2.550)
  GGT; Day 14, 24 h post dose | -1.96 (2.873) | -0.46 (4.187)

10. Primary Outcome: Part A: Change From Baseline in Creatinine, Bilirubin, and Total Bilirubin at the Indicated Time Points
Description: as for outcome 2
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles/Liter (micromol/L)
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
Micromoles/Liter (micromol/L)
  Creatinine; Day 7/Day 8, pre-dose | 2.31 (4.385) | -0.62 (5.104)
  Creatinine; Day 14, 24 h post dose | 3.64 (6.035) | 0.07 (3.259)
  Direct bilirubin; Day 7/Day 8, pre-dose | 0.33 (0.419) | 0.04 (0.398)
  Direct bilirubin; Day 14, 24 h post dose | 0.27 (0.496) | 0.10 (0.329)
  Total bilirubin; Day 7/Day 8, pre-dose | 1.23 (2.447) | 0.02 (2.590)
  Total bilirubin; Day 14, 24 h post dose | 0.90 (2.805) | 0.78 (1.720)

11. Primary Outcome: Part A: Change From Baseline in Calcium, Potassium, Sodium, Glucose, and Blood Urea Nitrogen (BUN) at the Indicated Time Points
Description: as for outcome 2
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
Millimoles per Liter (mmol/L)
  Calcium; Day 7/Day 8, pre-dose | 0.033 (0.0535) | 0.033 (0.0617)
  Calcium; Day 14, 24 h post dose | 0.033 (0.0850) | 0.029 (0.0588)
  Glucose; Day 7/Day 8, pre-dose | -0.053 (0.3333) | 0.012 (0.2888)
  Glucose; Day 14, 24 h post dose | 0.161 (0.2659) | 0.024 (0.4914)
  Potassium; Day 7/Day 8, pre-dose | 0.103 (0.2279) | 0.011 (0.3539)
  Potassium; Day 14, 24 h post dose | 0.161 (0.2562) | 0.065 (0.3347)
  Sodium; Day 7/Day 8, pre-dose | 1.21 (2.800) | 0.88 (1.560)
  Sodium; Day 14, 24 h post dose | 0.81 (1.297) | 0.83 (1.390)
  BUN; Day 7/Day 8, pre-dose | -0.530 (1.0830) | -0.192 (0.8124)
  BUN; Day 14, 24 h post dose | -0.464 (1.1979) | 0.111 (1.2147)

12. Primary Outcome: Part A: Number of Participants Meeting Criteria of Potential Clinical Importance for Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), and Heart Rate (HR) at Any Visit Post-Baseline
Description: Baseline was the Day 1 pre-dose measurement. Vital signs (SBP, DBP, and HR) were measured at Day 1 (30 minutes [min] and 6 h post-dose), Day 7 (pre-dose), and Day 14 (24 h post-dose). Potential clinical concern range for SBP was <85 millimeters of mercury (mmHg) (low) and >160 mmHg (high), for DBP <45 mmHg (low) and >100 mmHg (high) and for HR <40 bpm and >110 bpm. All measurements were obtained in supine position, after a 5-minute rest. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Day 1, Day 7, and Day 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
Participants
  SBP high | 1 | 1
  SBP low | 0 | 0
  DBP high | 0 | 0
  DBP low | 1 | 0
  HR high | 0 | 1
  HR low | 0 | 0

13. Primary Outcome: Part A: Number of Participants With Normal and Abnormal (Clinically Significant or Not Clinically Significant) Findings in 12-lead Electrocardiogram (ECG) at Any Visit Post-Baseline
Description: Baseline was the Day 1 (pre-dose) measurement. Single 12-lead ECGs were obtained using an ECG machine that automatically calculates the HR and measures PR, QRS, QT, and corrected QT intervals. Clinical significance was judged by the investigator. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Day 1, Day 7, and Day 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
Participants
  Normal | 2 | 13
  Abnormal - not clinically significant | 5 | 8
  Abnormal - clinically significant | 0 | 0

14. Primary Outcome: Part A: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) and Forced Vital Capacity (FVC) at the Indicated Time Points
Description: Baseline is Day 1 pre-dose. FEV1 and FVC are measures of lung function. FEV1 is defined as the maximal amount of air that can be forcefully exhaled in one second. FVC is defined as the maximum amount of air that can be forcibly blown out after a maximum inspiration. FEV1 and FVC measurements were repeated until three technically acceptable measurements (within 150 milliliters of each other) had been made. Only the best of three measurements were recorded. Baseline was the maximum of the planned pre-dose measurements on Day 1. Change from Baseline at any post-dose time point was calculated as the post-dose value minus the Baseline value. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Baseline (Day 1 [pre-dose]), Day 1 (1 h post-dose), Day 7 (pre-dose and 1 h post-dose), and Day 14 (24 h post-dose)
Population: Safety Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 7 | 21
Liters
  FEV1, Day 1, 1 h post dose | 0.15 [-0.01 to 0.30] | 0.10 [0.02 to 0.18]
  FEV1, Day 7/8, Pre-dose | 0.03 [-0.09 to 0.15] | -0.04 [-0.13 to 0.05]
  FEV1, Day 7/8, 1 h post dose | 0.27 [0.15 to 0.39] | 0.18 [0.10 to 0.26]
  FEV1, Day 14, 24 h post dose | -0.01 [-0.09 to 0.06] | 0.01 [-0.07 to 0.09]
  FVC, Day 1, 1 h post dose | 0.17 [-0.13 to 0.47] | 0.16 [0.01 to 0.32]
  FVC, Day 7/8, Predose | 0.02 [-0.23 to 0.26] | 0.00 [-0.12 to 0.13]
  FVC, Day 7/8, 1 h post dose | 0.33 [0.09 to 0.58] | 0.22 [0.09 to 0.36]
  FVC, Day 14, 24 h post dose | -0.04 [-0.30 to 0.22] | 0.10 [-0.07 to 0.27]

15. Primary Outcome: Part B: Adjusted Median Response of Cytokine (Interleukin 6 [IL6], Interleukin 8 [IL8], Tumor Necrosis Factor Alpha [TNFalpha]) Concentrations in Induced Sputum, on Day 7 and Day 14
Description: This outcome measure was used to estimate the inhibition levels of various doses of GSK2269557 by analyzing inflammatory cytokines IL6, IL8, and TNF alpha using Bayesian methods of statistical analysis, using non-informative prior distributions for all modeling parameters. Posterior medians (adjusted median response) and 95% credible intervals are reported here as medians and 95% confidence intervals respectively. 95% credible interval is reported as 2-sided 95% confidence in the statistical analyses. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Day 7 (pre-dose) and Day 14 (24 h post-dose)
Population: Safety Population
Measure: Median (95% Confidence Interval); unit: Picograms/milliliter (pg/mL)
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5 | 5
Picograms/milliliter (pg/mL)
  IL6, Day 7/Day 8 | 41.30 [22.07 to 78.24] | 37.40 [19.64 to 70.65] | 28.23 [14.80 to 53.18] | 30.82 [16.23 to 58.00] | 52.23 [28.73 to 94.94] | 31.25 [16.01 to 63.01] | 33.40 [17.52 to 63.23]
  IL6, Day 14 | 35.15 [17.72 to 70.01] | 37.60 [18.71 to 74.49] | 28.27 [14.10 to 56.22] | 22.68 [11.32 to 45.13] | 35.19 [18.32 to 66.93] | 42.56 [20.57 to 90.25] | 41.52 [20.62 to 82.81]
  IL8, Day 7/Day 8 | 2633.21 [1401.19 to 4879.27] | 2118.15 [1157.33 to 3866.74] | 1860.78 [995.35 to 3499.61] | 1523.63 [834.99 to 2745.90] | 2650.13 [1535.07 to 4634.07] | 2636.08 [1412.65 to 4978.59] | 2279.48 [1205.35 to 4210.75]
  IL8, Day 14 | 2942.28 [1375.08 to 6216.67] | 2664.75 [1269.52 to 5544.49] | 1879.92 [876.50 to 4056.53] | 1619.12 [778.39 to 3309.81] | 1356.35 [696.37 to 2645.82] | 2394.65 [1125.17 to 5196.20] | 2170.41 [1010.85 to 4582.03]
  TNFalpha, Day 7/Day 8 | 3.35 [1.22 to 8.98] | 1.55 [0.57 to 4.33] | 1.16 [0.42 to 3.25] | 1.54 [0.57 to 4.19] | 7.32 [3.02 to 17.85] | 3.68 [1.26 to 10.51] | 2.62 [0.94 to 7.15]
  TNFalpha, Day 14 | 2.91 [1.26 to 6.54] | 3.02 [1.33 to 7.00] | 1.25 [0.55 to 2.90] | 1.26 [0.55 to 2.87] | 3.99 [1.86 to 8.50] | 3.00 [1.34 to 6.75] | 1.53 [0.66 to 3.47]
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: GSK2269577 100 µg; Test type: Superiority or Other; p = 0.599, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.90, 95% CI 2-sided [0.39 to 2.07] — Comparison of IL6 concentrations at Day 7. This is the baseline corrected ratio of 100ug/placebo for day 7
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: GSK2269577 100 µg; Test type: Superiority or Other; p = 0.442, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 1.07, 95% CI 2-sided [0.43 to 2.59] — Comparison of IL6 concentrations at Day 14. This is the baseline corrected ratio of 100ug/placebo for day 14
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: GSK2269577 200 µg; Test type: Superiority or Other; p = 0.823, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.68, 95% CI 2-sided [0.30 to 1.57] — Comparison of IL6 concentrations at Day 7. This is the baseline corrected ratio of 200ug/placebo for day 7
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: GSK2269577 200 µg; Test type: Superiority or Other; p = 0.690, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 0.81, 95% CI 2-sided [0.33 to 1.97] — Comparison of IL6 concentrations at Day 14. This is the baseline corrected ratio of 200ug/placebo for day 14
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: GSK2269577 500 µg; Test type: Superiority or Other; p = 0.764, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.75, 95% CI 2-sided [0.33 to 1.71] — Comparison of IL6 concentrations at Day 7. This is the baseline corrected ratio of 500ug/placebo for day 7
Statistical Analysis 6: Comparison: Part B: Placebo vs Part B: GSK2269577 500 µg; Test type: Superiority or Other; p = 0.841, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 0.64, 95% CI 2-sided [0.27 to 1.56] — Comparison of IL6 concentrations at Day 14. This is the baseline corrected ratio of 500ug/placebo for day 14
Statistical Analysis 7: Comparison: Part B: Placebo vs Part B: GSK2269577 100 µg; Test type: Superiority or Other; p = 0.702, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.81, 95% CI 2-sided [0.35 to 1.81] — Comparison of IL8 concentrations at Day 7.This is the baseline corrected ratio of 100ug/placebo for day 7
Statistical Analysis 8: Comparison: Part B: Placebo vs Part B: GSK2269577 100 µg; Test type: Superiority or Other; p = 0.578, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 0.91, 95% CI 2-sided [0.33 to 2.47] — Comparison of IL8 concentrations at Day 14. This is the baseline corrected ratio of 100ug/placebo for day 14
Statistical Analysis 9: Comparison: Part B: Placebo vs Part B: GSK2269577 200 µg; Test type: Superiority or Other; p = 0.783, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.71, 95% CI 2-sided [0.29 to 1.70] — Comparison of IL8 concentrations at Day 7. This is the baseline corrected ratio of 200ug/placebo for day 7
Statistical Analysis 10: Comparison: Part B: Placebo vs Part B: GSK2269577 200 µg; Test type: Superiority or Other; p = 0.797, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 0.64, 95% CI 2-sided [0.22 to 1.87] — Comparison of IL8 concentrations at Day 14. This is the baseline corrected ratio of 200ug/placebo for day 14
Statistical Analysis 11: Comparison: Part B: Placebo vs Part B: GSK2269577 500 µg; Test type: Superiority or Other; p = 0.919, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.58, 95% CI 2-sided [0.27 to 1.26] — Comparison of IL8 concentrations at Day 7. This is the baseline corrected ratio of 500ug/placebo for day 7
Statistical Analysis 12: Comparison: Part B: Placebo vs Part B: GSK2269577 500 µg; Test type: Superiority or Other; p = 0.892, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 0.55, 95% CI 2-sided [0.21 to 1.43] — Comparison of IL8 concentrations at Day 14. This is the baseline corrected ratio of 500ug/placebo for day 14
Statistical Analysis 13: Comparison: Part B: Placebo vs Part B: GSK2269577 100 µg; Test type: Superiority or Other; p = 0.860, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.47, 95% CI 2-sided [0.11 to 1.93] — Comparison of TNFalpha concentrations at Day 7. This is the baseline corrected ratio of 100ug/placebo for day 7
Statistical Analysis 14: Comparison: Part B: Placebo vs Part B: GSK2269577 100 µg; Test type: Superiority or Other; p = 0.463, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 1.05, 95% CI 2-sided [0.38 to 2.86] — Comparison of TNFalpha concentrations at Day 14. This is the baseline corrected ratio of 100ug/placebo for day 14
Statistical Analysis 15: Comparison: Part B: Placebo vs Part B: GSK2269577 200 µg; Test type: Superiority or Other; p = 0.932, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.35, 95% CI 2-sided [0.09 to 1.42] — Comparison of TNFalpha concentrations at Day 7. This is the baseline corrected ratio of 200ug/placebo for day 7
Statistical Analysis 16: Comparison: Part B: Placebo vs Part B: GSK2269577 200 µg; Test type: Superiority or Other; p = 0.952, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 0.43, 95% CI 2-sided [0.16 to 1.17] — Comparison of TNFalpha concentrations at Day 14. This is the baseline corrected ratio of 200ug/placebo for day 14
Statistical Analysis 17: Comparison: Part B: Placebo vs Part B: GSK2269577 500 µg; Test type: Superiority or Other; p = 0.873, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.46, 95% CI 2-sided [0.12 to 1.81] — Comparison of TNFalpha concentrations at Day 7. This is the baseline corrected ratio of 500ug/placebo for day 7
Statistical Analysis 18: Comparison: Part B: Placebo vs Part B: GSK2269577 500 µg; Test type: Superiority or Other; p = 0.953, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 0.43, 95% CI 2-sided [0.16 to 1.16] — Comparison of TNFalpha concentrations at Day 14. This is the baseline corrected ratio of 500ug/placebo for day 14
Statistical Analysis 19: Comparison: Part B: Placebo vs Part B: GSK2269577 700 µg; Test type: Superiority or Other; p = 0.281, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio9 = 1.26, 95% CI 2-sided [0.56 to 2.82] — Comparison of IL6 concentrations at Day 7. This is the baseline corrected ratio of 700ug/placebo for day 7
Statistical Analysis 20: Comparison: Part B: Placebo vs Part B: GSK2269577 700 µg; Test type: Superiority or Other; p = 0.500, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 1.00, 95% CI 2-sided [0.42 to 2.35] — Comparison of IL6 concentrations at Day 14. This is the baseline corrected ratio of 700ug/placebo for day 14
Statistical Analysis 21: Comparison: Part B: Placebo vs Part B: GSK2269577 1000 µg; Test type: Superiority or Other; p = 0.744, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.76, 95% CI 2-sided [0.32 to 1.77] — Comparison of IL6 concentrations at Day 7. This is the baseline corrected ratio of 1000ug/placebo for day 7
Statistical Analysis 22: Comparison: Part B: Placebo vs Part B: GSK2269577 1000 µg; Test type: Superiority or Other; p = 0.334, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 1.21, 95% CI 2-sided [0.49 to 3.04] — Comparison of IL6 concentrations at Day 14. This is the baseline corrected ratio of 1000ug/placebo for day 14
Statistical Analysis 23: Comparison: Part B: Placebo vs Part B: GSK2269577 2000 µg; Test type: Superiority or Other; p = 0.698, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.81, 95% CI 2-sided [0.35 to 1.85] — Comparison of IL6 concentrations at Day 7. This is the baseline corrected ratio of 2000ug/placebo for day 7
Statistical Analysis 24: Comparison: Part B: Placebo vs Part B: GSK2269577 2000 µg; Test type: Superiority or Other; p = 0.353, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 1.18, 95% CI 2-sided [0.48 to 2.88] — Comparison of IL6 concentrations at Day 14. This is the baseline corrected ratio of 2000ug/placebo for day 14
Statistical Analysis 25: Comparison: Part B: Placebo vs Part B: GSK2269577 700 µg; Test type: Superiority or Other; p = 0.489, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio9 = 1.01, 95% CI 2-sided [0.45 to 2.26] — Comparison of IL8 concentrations at Day 7. This is the baseline corrected ratio of 700ug/placebo for day 7
Statistical Analysis 26: Comparison: Part B: Placebo vs Part B: GSK2269577 700 µg; Test type: Superiority or Other; p = 0.940, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 0.46, 95% CI 2-sided [0.17 to 1.23] — Comparison of IL8 concentrations at Day 14. This is the baseline corrected ratio of 700ug/placebo for day 14
Statistical Analysis 27: Comparison: Part B: Placebo vs Part B: GSK2269577 1000 µg; Test type: Superiority or Other; p = 0.495, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 1.01, 95% CI 2-sided [0.42 to 2.40] — Comparison of IL8 concentrations at Day 7. This is the baseline corrected ratio of 1000ug/placebo for day 7
Statistical Analysis 28: Comparison: Part B: Placebo vs Part B: GSK2269577 1000 µg; Test type: Superiority or Other; p = 0.647, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 0.82, 95% CI 2-sided [0.28 to 2.37] — Comparison of IL8 concentrations at Day 14. This is the baseline corrected ratio of 1000ug/placebo for day 14
Statistical Analysis 29: Comparison: Part B: Placebo vs Part B: GSK2269577 2000 µg; Test type: Superiority or Other; p = 0.646, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.87, 95% CI 2-sided [0.40 to 1.86] — Comparison of IL8 concentrations at Day 7. This is the baseline corrected ratio of 2000ug/placebo for day 7
Statistical Analysis 30: Comparison: Part B: Placebo vs Part B: GSK2269577 2000 µg; Test type: Superiority or Other; p = 0.741, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 0.74, 95% CI 2-sided [0.29 to 1.90] — Comparison of IL8 concentrations at Day 14. This is the baseline corrected ratio of 2000ug/placebo for day 14
Statistical Analysis 31: Comparison: Part B: Placebo vs Part B: GSK2269577 700 µg; Test type: Superiority or Other; p = 0.109, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio9 = 2.18, 95% CI 2-sided [0.62 to 7.95] — Comparison of TNFalpha concentrations at Day 7. This is the baseline corrected ratio of 700ug/placebo for day 7
Statistical Analysis 32: Comparison: Part B: Placebo vs Part B: GSK2269577 700 µg; Test type: Superiority or Other; p = 0.240, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 1.37, 95% CI 2-sided [0.55 to 3.45] — Comparison of TNFalpha concentrations at Day 14. This is the baseline corrected ratio of 700ug/placebo for day 14
Statistical Analysis 33: Comparison: Part B: Placebo vs Part B: GSK2269577 1000 µg; Test type: Superiority or Other; p = 0.447, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 1.10, 95% CI 2-sided [0.27 to 4.44] — Comparison of TNFalpha concentrations at Day 7. This is the baseline corrected ratio of 1000ug/placebo for day 7
Statistical Analysis 34: Comparison: Part B: Placebo vs Part B: GSK2269577 1000 µg; Test type: Superiority or Other; p = 0.472, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 1.03, 95% CI 2-sided [0.39 to 2.74] — Comparison of TNFalpha concentrations at Day 14. This is the baseline corrected ratio of 1000ug/placebo for day 14
Statistical Analysis 35: Comparison: Part B: Placebo vs Part B: GSK2269577 2000 µg; Test type: Superiority or Other; p = 0.698, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 7; Adjusted Median Ratio = 0.78, 95% CI 2-sided [0.21 to 2.90] — Comparison of TNFalpha concentrations at Day 7. This is the baseline corrected ratio of 2000ug/placebo for day 7
Statistical Analysis 36: Comparison: Part B: Placebo vs Part B: GSK2269577 2000 µg; Test type: Superiority or Other; p = 0.911, Bayesian repeated measures — Posterior Probability the True Treatment Ratio <1 for Day 14; Adjusted Median Ratio = 0.53, 95% CI 2-sided [0.21 to 1.37] — Comparison of TNFalpha concentrations at Day 14. This is the baseline corrected ratio of 2000ug/placebo for day 14

16. Secondary Outcome: Part A: Day 1 Plasma Concentration of GSK2269577 up to 6 Hours Post Dose
Description: A 2 mL blood sample for pharmacokinetic (PK) analysis was collected at each of the indicated time point. Only those participants who were available at the indicated time points were analyzed (represented by n=X in the category titles). A value of NA indicates that the geometric mean or 95% confidence interval is not available.
Time Frame: Day 1 (Pre-dose, 5 min, 30 min, 1, 2, 4 & 6 hours post-dose)
Population: PK Population: participants in the Safety Population for whom a PK sample was obtained and analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 21
pg/mL
  Pre-dose; n=0 | NA [NA to NA] — A value of NA indicates that the geometric mean or 95% confidence interval is not available.
  5 min; n=21 | 386.2 [287.5 to 518.7]
  30 min; n=21 | 337.2 [274.6 to 414.0]
  1 h; n=21 | 379.1 [320.2 to 448.9]
  2 h; n=21 | 531.1 [448.2 to 629.4]
  4 h; n=21 | 419.5 [357.6 to 492.1]
  6 h; n=21 | 334.4 [287.0 to 389.6]

17. Secondary Outcome: Part B: Day 1 Plasma Concentration of GSK2269577 up to 6 Hours Post Dose
Description: A 2 mL blood sample for pharmacokinetic (PK) analysis was collected at each of the indicated time point. Concentration measurements were log-transformed. Only those participants who were available at the indicated time points were analyzed (represented by n=X,X in the category titles). A value of NA indicates that the geometric mean or 95% confidence interval is not available.
Time Frame: Pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, and 6 h post-dose on Day 1
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 5
pg/mL
  Pre-dose; n=0,0,0,0,0,0 | NA [NA to NA] — A value of NA indicates that the geometric mean or 95% confidence interval is not available. | NA [NA to NA] — A value of NA indicates that the geometric mean or 95% confidence interval is not available. | NA [NA to NA] — A value of NA indicates that the geometric mean or 95% confidence interval is not available. | NA [NA to NA] — A value of NA indicates that the geometric mean or 95% confidence interval is not available. | NA [NA to NA] — A value of NA indicates that the geometric mean or 95% confidence interval is not available. | NA [NA to NA] — A value of NA indicates that the geometric mean or 95% confidence interval is not available.
  5 min; n=5,5,5,6,5,5 | 55.3 [33.7 to 90.7] | 80.4 [38.4 to 168.2] | 173.1 [88.4 to 339.0] | 466.6 [147.3 to 1478.0] | 853.4 [380.2 to 1915.6] | 982.9 [311.1 to 3105.3]
  30 min; n=5,5,5,6,5,5 | 51.7 [36.2 to 74.1] | 73.8 [41.6 to 130.8] | 203 [111.2 to 370.5] | 402.3 [218.0 to 742.5] | 556.9 [384.8 to 806.0] | 1011.6 [757.1 to 1351.6]
  1 h; n=5,5,5,6,5,5 | 61.3 [45.7 to 82.3] | 77.2 [44.1 to 135.2] | 253.2 [155.0 to 413.8] | 429.1 [294.2 to 626.0] | 599.7 [370.5 to 970.7] | 1203.3 [799.1 to 1812.0]
  2 h; n=5,5,5,6,5,5 | 60.6 [44.8 to 81.9] | 88.8 [60.2 to 130.9] | 300.9 [173.7 to 521.1] | 556.7 [372.4 to 832.3] | 672.3 [434.0 to 1041.5] | 1402 [892.8 to 2201.4]
  4 h; n=5,5,5,6,5,5 | 45.0 [33.1 to 61.2] | 73.4 [60.5 to 89.1] | 251 [146.0 to 431.6] | 391.6 [303.3 to 505.5] | 468.7 [305.5 to 719.2] | 1098.5 [781.9 to 1543.2]
  6 h; n=5,5,5,6,5,5 | 38.3 [29.7 to 49.5] | 63.8 [50.7 to 80.3] | 201.5 [128.3 to 316.6] | 294.6 [222.3 to 390.4] | 466.5 [273.1 to 796.6] | 900.8 [723.8 to 1121.0]

18. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of GSK2269577 on Day 7
Description: Blood samples were collected to determine the plasma concentrations of GSK2269577 immediately after dosing on Day 7. Day 7 sampling could be done on Day 7 or Day 8.
Time Frame: Day 7 immediately after dosing
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 21
pg/mL | 1109.1 [901.5 to 1364.5]

19. Secondary Outcome: Part B: Maximum Observed Plasma Concentration (Cmax) of GSK2269577 on Day 7
Description: Blood samples were collected to determine the plasma concentrations of GSK2269577 immediately after dosing on Day 7. Concentration values were log-transformed. Day 7 sampling could be done on Day 7 or Day 8.
Time Frame: Day 7 immediately after dosing
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 5
pg/mL | 109.6 [62.6 to 191.8] | 203.4 [140.3 to 294.8] | 511.8 [233.2 to 1123.3] | 1022.2 [623.7 to 1675.2] | 1655.1 [803.2 to 3410.4] | 2923.4 [1769.4 to 4830.0]

20. Secondary Outcome: Part A: Trough Concentration (Ctau) of GSK2269577 on Day 7 and Day 15
Description: Blood samples were collected to determine the (trough) plasma concentration of GSK2269577 on Day 7 (pre-dose) and Day 15 (24 hours after dosing on Day 14). Day 7 assessments could be done either on Day 7 or on Day 8.
Time Frame: Day 7 and Day 15
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Part A: GSK2269577 1000 µg
Number analyzed (Participants) | 21
pg/mL
  Day 7/Day 8 | 604.1 [496.6 to 735.0]
  Day 15 | 711.2 [561.8 to 900.3]

21. Secondary Outcome: Part B: Trough Concentration (Ctau) of GSK2269577 on Day 7 and Day 15
Description: as for outcome 20
Time Frame: Day 7 and Day 15
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 6 | 5 | 5
pg/mL
  Day 7/Day 8 | 55.3 [41.22 to 74.21] | 119.17 [78.47 to 180.97] | 314.38 [182.64 to 541.16] | 588.09 [486.63 to 710.69] | 724.33 [581.37 to 902.45] | 1468.94 [1000.50 to 2156.70]
  Day 15 | 74.93 [48.26 to 116.33] | 128.71 [92.02 to 180.03] | 237.36 [66.38 to 848.74] | 665.9 [497.61 to 891.10] | 1218.5 [985.88 to 1506.01] | 1767.34 [1079.72 to 2892.86]

22. Secondary Outcome: Part B: Number of Times Rescue Medication Was Used by Participants Daily, During the Treatment Period
Description: Rescue medication was identified from concomitant medication records and the patient diaries which were provided to the participants to record data throughout the treatment period. Only participants who used rescue medication were analyzed. The value NA indicates that the standard deviation could not be calculated as only one participant was analyzed.
Time Frame: Day 1 to Day 15
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Number of times
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 3 | 1 | 1 | 0 | 1 | 3 | 1
Number of times | 2.00 (0.00) | 2.3 (NA) — The value NA indicates that the standard deviation could not be calculated as only one participant was analyzed. | 2.2 (NA) — The value NA indicates that the standard deviation could not be calculated as only one participant was analyzed. |  | 1.0 (NA) — The value NA indicates that the standard deviation could not be calculated as only one participant was analyzed. | 1.4 (0.63) | 1.0 (NA) — The value NA indicates that the standard deviation could not be calculated as only one participant was analyzed.

23. Secondary Outcome: Part B: Number of Participants With at Least One Non-serious Adverse Event (AE), Serious Adverse Event (SAE), or Drug-related Adverse Event
Description: as for outcome 1
Time Frame: From the start of study treatment until follow-up (assessed for approximately 19 days)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5 | 5
Participants
  At least one AE | 3 | 3 | 2 | 1 | 3 | 4 | 2
  At least one SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  At least one drug-related AE | 0 | 0 | 1 | 0 | 3 | 4 | 2

24. Secondary Outcome: Part B: Change From Baseline in Counts of Basophils, Eosinophils, Lymphocytes, Monocytes, Platelets, White Blood Cells (WBC), Total Neutrophils (Total ANC) at the Indicated Time Points
Description: Blood samples were collected for measurement for the indicated tests. Change from Baseline at any post-dose visit was calculated as the post-dose visit value minus the Baseline value. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5 | 5
10^9 cells per liter (GI/L)
  Basophils; Day 7/Day 8, pre-dose | 0.014 (0.0241) | -0.002 (0.0228) | 0.01 (0.0187) | 0.004 (0.0182) | 0.007 (0.0052) | -0.005 (0.01) | 0 (0.01)
  Basophils; Day 14, 24 h post dose | 0.004 (0.0167) | -0.006 (0.0261) | 0.01 (0.0122) | -0.002 (0.0192) | 0.007 (0.0175) | -0.008 (0.0189) | 0.01 (0.0122)
  Eosinophils; Day 7/Day 8, pre-dose | -0.002 (0.0576) | 0.01 (0.0485) | -0.034 (0.0702) | -0.026 (0.0498) | 0.022 (0.1289) | -0.002 (0.0287) | 0.012 (0.0438)
  Eosinophils; Day 14, 24 h post dose | 0.046 (0.0472) | -0.01 (0.0292) | -0.046 (0.0378) | -0.054 (0.1498) | 0.025 (0.1078) | 0.023 (0.0222) | 0.022 (0.0396)
  Lymphocytes; Day 7/Day 8, pre-dose | 0.242 (0.4797) | -0.178 (0.5657) | -0.022 (0.1326) | -0.094 (0.3092) | 0.093 (0.2813) | -0.118 (0.3223) | -0.218 (0.6236)
  Lymphocytes; Day 14, 24 h post dose | -0.09 (0.4499) | -0.264 (0.3134) | -0.216 (0.208) | 0.092 (0.9722) | 0.21 (0.3855) | -0.243 (0.3054) | -0.398 (0.736)
  Monocytes; Day 7/Day 8, pre-dose | -0.062 (0.0867) | 0.05 (0.0941) | -0.02 (0.0806) | 0.05 (0.2108) | 0.018 (0.1209) | 0.165 (0.5166) | -0.08 (0.1398)
  Monocytes; Day 14, 24 h post dose | -0.022 (0.0676) | -0.012 (0.0926) | -0.036 (0.0829) | -0.004 (0.1313) | 0.03 (0.0699) | 0.108 (0.3437) | -0.11 (0.0834)
  Platelets; Day 7/Day 8, pre-dose | -13.8 (14.22) | -0.8 (18.07) | 10 (24.52) | 15.6 (17.78) | 11.7 (15.41) | 26.5 (32.77) | -0.6 (14.4)
  Platelets; Day 14, 24 h post dose | -3.3 (22.25) | -13 (26.52) | -7.2 (20.41) | -1.4 (44.86) | 7 (19.81) | -8.3 (51.57) | -11.4 (29.39)
  WBC; Day 7/Day 8, pre-dose | 0.372 (1.5852) | -0.024 (1.1519) | 0.102 (1.1107) | 0.926 (3.1314) | 0.497 (0.8673) | 0.5 (2.676) | -0.802 (0.7889)
  WBC; Day 14, 24 h post dose | -0.49 (0.5204) | -0.864 (1.4151) | -0.164 (0.7907) | -0.178 (2.2899) | 0.648 (1.143) | 0.825 (1.6016) | -1.012 (1.3388)
  Total ANC; Day 7/Day 8, pre-dose | 0.164 (0.9782) | 0.09 (0.6553) | 0.17 (1.0481) | 1.018 (2.6669) | 0.335 (0.5921) | 0.448 (2.153) | -0.51 (0.285)
  Total ANC; Day 14, 24 h post dose | -0.44 (0.4288) | -0.538 (1.1027) | 0.134 (0.801) | -0.18 (1.469) | 0.385 (1.2151) | 0.958 (1.8925) | -0.51 (0.7931)

25. Secondary Outcome: Part B: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) at the Indicated Time Points
Description: Blood samples were collected for measurement for the indicated tests. MCHC is one of the red blood cell (RBC) indices. Change from Baseline at any post-dose visit was calculated as the post-dose visit value minus the Baseline value. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5 | 5
g/L
  Hemoglobin; Day 7/Day 8, pre-dose | 3 (2.55) [lower limit 2.55] | 0.8 (5.76) | 3.8 (6.76) | 1 (4.74) | 0.3 (5.65) | 6 (5.89) | 1 (3.39)
  Hemoglobin; Day 14, 24 h post dose | 4.2 (6.14) [lower limit 6.14] | -1.2 (6.14) | -0.6 (8.02) | -2 (6.86) | -2.2 (2.14) | -0.3 (4.65) | -0.2 (4.44)
  MCHC; Day 7/Day 8, pre-dose | -2.4 (2.07) [lower limit 2.07] | -0.6 (8.17) | -4.0 (7.31) | -4.4 (9.61) | 0.5 (5.17) | 3.3 (8.18) | 7.8 (10.85)
  MCHC; Day 14, 24 h post dose | 3.8 (5.07) [lower limit 5.07] | -2.6 (3.51) | -4.4 (8.73) | 3.0 (4.00) | 2.5 (3.83) | -8.5 (7.59) | 1.6 (11.76)

26. Secondary Outcome: Part B: Change From Baseline in Counts of RBCs and Reticulocytes at the Indicated Time Points
Description: as for outcome 24
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/Liter (TI/L)
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 4 | 5
10^12 cells/Liter (TI/L)
  RBC; Day 7/Day 8, pre-dose | 0.076 (0.1148) | 0.036 (0.1549) | 0.18 (0.2703) | 0.058 (0.1314) | -0.023 (0.1508) | 0.14 (0.0879) | -0.058 (0.1252)
  RBC; Day 14, 24 h post dose | 0.11 (0.1891) | -0.038 (0.1663) | 0.034 (0.1785) | -0.07 (0.1815) | -0.083 (0.0958) | 0.042 (0.1031) | -0.084 (0.1496)
  Reticulocytes; Day 7/Day 8, pre-dose | -0.00064 (0.01328) | 0.00714 (0.020838) | 0.01298 (0.011129) | 0.01258 (0.014565) | 0.00397 (0.008856) | 0.00882 (0.018576) | 0.01792 (0.012824)
  Reticulocytes; Day 14, 24 h post dose | 0.0034 (0.014934) | 0.0006 (0.010183) | 0.01032 (0.015404) | 0.0156 (0.013092) | -0.00172 (0.005382) | -0.01063 (0.018329) | 0.00884 (0.015546)

27. Secondary Outcome: Part B: Change From Baseline in Hematocrit at the Indicated Time Points
Description: as for outcome 24
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5 | 5
Ratio
  Day 7/Day 8, pre-dose | 0.012 (0.0084) | 0.004 (0.0182) | 0.018 (0.0259) | 0.01 (0.01) | 0 (0.0141) | 0.015 (0.0058) | -0.010 (0.0235)
  Day 14, 24 h post dose | 0.008 (0.0217) | 0 (0.0212) | 0.006 (0.0152) | -0.012 (0.0217) | -0.01 (0.0063) | 0.01 (0.0082) | -0.004 (0.0207)

28. Secondary Outcome: Part B: Change From Baseline in Mean Corpuscle Hemoglobin (MCH) at the Indicated Time Points
Description: Blood samples were collected for measurement for the indicated tests. MCH is one of the red blood cell indices. Change from Baseline at any post-dose visit was calculated as the post-dose visit value minus the Baseline value. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 4 | 5
pg
  Day 7/Day 8, pre-dose | 0.18 (0.415) | -0.06 (0.397) | -0.36 (0.351) | -0.08 (0.669) | 0.2 (0.529) | 0.35 (0.961) | 0.58 (0.46)
  Day 14, 24 h post dose | 0.18 (0.626) | 0.02 (0.259) | -0.34 (0.74) | 0.12 (0.396) | 0.1 (0.363) | -0.33 (0.754) | 0.52 (0.268)

29. Secondary Outcome: Part B: Change From Baseline in Mean Corpuscle Volume (MCV) at the Indicated Time Points
Description: Blood samples were collected for measurement for the indicated tests. MCV is one of the RBC indices. Change from Baseline at any post-dose visit was calculated as the post-dose visit value minus the Baseline value. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 4 | 5
fL
  MCV; Day 7/Day 8, pre-dose | 1.24 (0.706) | -0.14 (1.794) | -0.12 (1.708) | 0.88 (1.085) | 0.42 (2.302) | 0.20 (0.583) | -0.70 (2.719)
  MCV; Day 14, 24 h post dose | -0.66 (1.537) | 0.80 (1.257) | 0.26 (1.935) | -0.62 (1.281) | -0.53 (1.601) | 1.53 (0.699) | 0.98 (3.155)

30. Secondary Outcome: Part B: Change From Baseline in Albumin and Total Protein at the Indicated Time Points
Description: as for outcome 24
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5 | 5
g/L
  Albumin; Day 7/Day 8, pre-dose | 0.96 (1.773) | 1.22 (1.571) | 0.96 (3.012) | 0.88 (0.887) | -0.6 (1.814) | 1.18 (1.069) | 0.3 (1.49)
  Albumin; Day 14, 24 h post dose | 0.9 (2.965) | 0.7 (2.134) | -0.12 (2.538) | -1.16 (2.157) | -1.13 (1.365) | 0.44 (1.001) | 0.26 (1.187)
  Total protein; Day 7/Day 8, pre-dose | 1.34 (2.46) | 0.72 (1.203) | 2.22 (4.953) | 0.98 (2.039) | -1.4 (2.662) | 1.78 (2.338) | 1.12 (1.571)
  Total protein; Day 14, 24 h post dose | 0.96 (3.392) | 0.96 (2.393) | -0.16 (3.737) | -1.96 (3.635) | -2.13 (2.156) | 0.72 (1.154) | 0.7 (2.277)

31. Secondary Outcome: Part B: Change From Baseline in Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), and Gamma Glutamyl Transferase (GGT) at the Indicated Time Points
Description: as for outcome 24
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5 | 5
International Units per Liter (IU/L)
  ALP; Day 7/Day 8, pre-dose | 1.88 (5.45) | 1.62 (5.756) | 1.64 (7.946) | 5.7 (9.986) | -0.95 (7.807) | -0.92 (22.572) | 1.66 (5.465)
  ALP; Day 14, 24 h post dose | 1.54 (4.503) | 4.78 (7.294) | -0.2 (6.109) | 0.26 (9.829) | -1.1 (8.535) | -5.34 (19.016) | 5.2 (4.038)
  ALT; Day 7/Day 8, pre-dose | 1.58 (2.24) | 3.66 (6.057) | -2.44 (7.23) | 2.6 (4.994) | -0.1 (2.994) | -2.4 (5.036) | 1.42 (2.791)
  ALT; Day 14, 24 h post dose | 0.36 (2.268) | 2.18 (3.17) | -2.76 (6.176) | 0.84 (5.223) | -0.72 (4.63) | -2.86 (5.478) | 1.58 (3.754)
  AST; Day 7/Day 8, pre-dose | 1.38 (2.464) | 3.76 (11.142) | -0.42 (3.13) | 0.26 (5.185) | -0.22 (3.672) | -2.56 (5.607) | 3.04 (2.048)
  AST; Day 14, 24 h post dose | 0.44 (1.691) | 0.16 (1.673) | -2.44 (3.443) | -1.64 (6.027) | 0.02 (3.129) | -1.66 (4.536) | 2.66 (1.25)
  GGT; Day 7/Day 8, pre-dose | -0.6 (2.119) | -0.3 (1.856) | -0.96 (4.556) | -0.3 (4.471) | 1.88 (4.747) | -3.18 (9.7) | 0.74 (1.141)
  GGT; Day 14, 24 h post dose | -0.64 (0.934) | 0.1 (2.625) | -2.64 (6.532) | -0.72 (5.485) | 1.52 (5.783) | -6.16 (17.113) | 0.54 (1.923)

32. Secondary Outcome: Part B: Change From Baseline in Creatinine, Bilirubin, and Total Bilirubin at the Indicated Time Points
Description: as for outcome 24
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles/Liter (micromol/L)
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5 | 5
Micromoles/Liter (micromol/L)
  Direct bilirubin; Day 7/Day 8, pre-dose | -0.02 (0.327) | 0.24 (0.493) | -0.28 (0.881) | 0.16 (0.261) | 0.23 (0.65) | -0.18 (1.36) | -0.32 (0.37)
  Direct bilirubin; Day 14, 24 h post dose | -0.1 (0.453) | -0.02 (0.192) | -0.58 (0.581) | 0.22 (0.409) | 0.2 (0.429) | 0.02 (0.554) | -0.14 (0.456)
  Total bilirubin; Day 7/Day 8, pre-dose | 0.28 (2.255) | 0.56 (2.151) | -0.7 (4.049) | 0.72 (2.196) | 1.08 (2.775) | -0.86 (1.75) | -1.5 (1.739)
  Total bilirubin; Day 14, 24 h post dose | -0.5 (3.389) | 0.08 (0.87) | -2.08 (2.387) | 0.52 (2.7) | 1.22 (3.008) | 0.5 (2.804) | -1.06 (1.479)
  Creatinine; Day 7/Day 8, pre-dose | 4.52 (4.533) | 1.6 (3.77) | 4.38 (2.217) | -0.3 (4.567) | 0.52 (4.397) | 3.48 (3.084) | 0.76 (5.421)
  Creatinine; Day 14, 24 h post dose | 1.58 (7.276) | 0.76 (3.319) | 4.84 (4.636) | -0.46 (6.98) | 2.05 (3.17) | 1.36 (2.545) | 1.42 (5.058)

33. Secondary Outcome: Part B: Change From Baseline in Calcium, Potassium, Sodium, Glucose, and Blood Urea Nitrogen (BUN) at the Indicated Time Points
Description: as for outcome 24
Time Frame: Baseline (Day 1 [pre-dose]), Day 7 (pre-dose), and Day 14 (24 hours [h] post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5 | 5
Millimoles per Liter (mmol/L)
  Calcium; Day 7/Day 8, pre-dose | 0.048 (0.0444) | 0.044 (0.0397) | 0.06 (0.0579) | 0.01 (0.0648) | -0.008 (0.0655) | 0.066 (0.0811) | 0.044 (0.0365)
  Calcium; Day 14, 24 h post dose | 0.024 (0.0865) | -0.012 (0.0482) | 0.05 (0.0696) | -0.01 (0.0758) | -0.042 (0.0422) | 0.03 (0.0292) | 0.036 (0.0568)
  Glucose; Day 7/Day 8, pre-dose | -0.06 (0.2939) | 0.054 (0.4057) | 0.05 (0.1937) | -0.43 (1.4084) | -0.11 (0.5658) | 0.11 (0.4369) | -0.246 (0.273)
  Glucose; Day 14, 24 h post dose | -0.086 (0.3743) | -0.142 (0.3746) | 0.26 (0.5456) | 0.054 (0.2294) | -0.34 (0.7332) | -0.076 (0.3518) | -0.314 (0.3871)
  Potassium; Day 7/Day 8, pre-dose | 0.246 (0.3088) | 0.09 (0.2793) | 0.434 (0.5451) | -0.204 (0.2563) | 0.135 (0.3172) | 0.276 (0.3566) | 0.192 (0.4587)
  Potassium; Day 14, 24 h post dose | 0.19 (0.1944) | 0.12 (0.4282) | 0.336 (0.5268) | -0.128 (0.3241) | 0.013 (0.203) | 0.14 (0.1259) | 0.072 (0.5946)
  Sodium; Day 7/Day 8, pre-dose | 0 (1.206) | 0.6 (1.626) | -0.12 (1.714) | 1.18 (1.139) | -0.33 (2.072) | 0.7 (1.815) | -0.84 (2.137)
  Sodium; Day 14, 24 h post dose | -0.16 (1.301) | -0.04 (3.233) | 0.58 (1.399) | 0.46 (1.447) | -0.18 (2.515) | 1.06 (1.074) | -0.4 (2.72)
  Urea/BUN; Day 7/Day 8, pre-dose | 0.314 (0.7077) | -0.504 (0.6955) | 0.342 (0.8193) | -0.91 (1.0653) | -0.29 (0.4396) | -0.244 (1.2909) | 0.162 (1.2285)
  Urea/BUN; Day 14, 24 h post dose | -0.232 (0.3592) | -0.124 (0.7502) | 0.142 (1.0269) | -0.906 (1.6431) | -0.335 (0.2793) | -0.364 (0.8554) | 0.186 (2.0478)

34. Secondary Outcome: Part B: Number of Participants Meeting Criteria of Potential Clinical Importance for Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), and Heart Rate (HR) at Any Visit Post-Baseline
Description: Baseline was the Day 1 pre-dose measurement. Vital signs (SBP, DBP, and HR) were measured at Day 1 (30 minutes [min] and 6 h post-dose), Day 7 (pre-dose), and Day 14 (24 h post-dose). All measurements were obtained in supine position, after a 5-minute rest. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Day 1, Day 7, and Day 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5 | 5
Participants
  SBP high | 0 | 0 | 1 | 1 | 1 | 0 | 0
  SBP low | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP high | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP low | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HR high | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HR low | 0 | 0 | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Part B: Number of Participants With Normal and Abnormal (Clinically Significant or Not Clinically Significant) Findings in 12-lead Electrocardiogram (ECG) at Any Visit Post-Baseline
Description: Baseline was the Day 1 (pre-dose) measurement. Single 12-lead ECGs were obtained using an ECG machine that automatically calculates the HR and measures PR, QRS, QT, and corrected QT intervals. Day 7 assessments could be conducted on Day 7 or Day 8.
Time Frame: Day 1, Day 7, and Day 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5 | 5
Participants
  Normal | 4 | 5 | 3 | 2 | 5 | 5 | 4
  Abnormal - not clinically significant | 1 | 0 | 2 | 3 | 1 | 0 | 1
  Abnormal - clinically significant | 0 | 0 | 0 | 0 | 0 | 0 | 0

36. Secondary Outcome: Part B: Forced Expiratory Volume in One Second (FEV1) and Forced Vital Capacity (FVC) at Screening and Follow-up
Description: FEV1 and FVC are measures of lung function. FEV1 is defined as the maximal amount of air that can be forcefully exhaled in one second. FVC is defined as the maximum amount of air that can be forcibly blown out after a maximum inspiration. FEV1 and FVC measurements were repeated until three technically acceptable measurements (within 150 milliliters of each other) had been made. Only the best of three measurements were recorded.
Time Frame: Screening (up to 30 days prior to Day 1) and Follow-up (approximately Day 19)
Population: Safety Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 6 | 5 | 5
Liters
  FEV1, Screening | 1.586 [1.093 to 2.079] | 1.387 [0.783 to 1.99] | 1.533 [0.784 to 2.282] | 1.558 [0.916 to 2.199] | 1.573 [1.092 to 2.055] | 1.36 [1.126 to 1.594] | 1.407 [0.768 to 2.046]
  FEV1, Follow-up | 1.494 [1.174 to 1.813] | 1.272 [0.69 to 1.855] | 1.523 [0.775 to 2.271] | 1.34 [1.092 to 1.589] | 1.501 [0.989 to 2.013] | 1.405 [0.948 to 1.861] | 1.431 [0.834 to 2.028]
  FVC, Screening | 3.05 [2.476 to 3.624] | 3.08 [1.901 to 4.259] | 3.632 [2.585 to 4.679] | 4.348 [3.565 to 5.131] | 3.277 [2.389 to 4.164] | 2.958 [1.6 to 4.316] | 3.156 [2.099 to 4.213]
  FVC, Follow-up | 2.96 [2.432 to 3.488] | 3.042 [1.809 to 4.275] | 3.764 [2.533 to 4.995] | 4.192 [3.527 to 4.857] | 3.137 [2.057 to 4.217] | 3.03 [1.691 to 4.369] | 3.192 [1.968 to 4.416]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs), defined as those events occurring from the start of treatment until follow-up (up to approximately 19 days), are reported.
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all participants who received at least one dose of study treatment.
Arm/Group | Part A: Placebo | Part A: GSK2269577 1000 µg | Part B: Placebo | Part B: GSK2269577 100 µg | Part B: GSK2269577 200 µg | Part B: GSK2269577 500 µg | Part B: GSK2269577 700 µg | Part B: GSK2269577 1000 µg | Part B: GSK2269577 2000 µg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/21 | 0/5 | 0/5 | 0/5 | 0/5 | 0/6 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/21 | 0/5 | 0/5 | 0/5 | 0/5 | 0/6 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/7 | 7/21 | 3/5 | 3/5 | 2/5 | 1/5 | 3/6 | 4/5 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=7) | Part A: GSK2269577 1000 µg (N=21) | Part B: Placebo (N=5) | Part B: GSK2269577 100 µg (N=5) | Part B: GSK2269577 200 µg (N=5) | Part B: GSK2269577 500 µg (N=5) | Part B: GSK2269577 700 µg (N=6) | Part B: GSK2269577 1000 µg (N=5) | Part B: GSK2269577 2000 µg (N=5)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=7) | Part A: GSK2269577 1000 µg (N=21) | Part B: Placebo (N=5) | Part B: GSK2269577 100 µg (N=5) | Part B: GSK2269577 200 µg (N=5) | Part B: GSK2269577 500 µg (N=5) | Part B: GSK2269577 700 µg (N=6) | Part B: GSK2269577 1000 µg (N=5) | Part B: GSK2269577 2000 µg (N=5)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0 | 1 | 0 | 3 | 4 | 2
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 (0) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.